CLINICAL TRIAL: NCT02959658
Title: Dimethyl Fumarate Treatment of Primary Progressive Multiple Sclerosis
Acronym: FUMAPMS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Biogen (Industry)
Responsible Party: Principal Investigator, Jacob L Talbot, Principal Investigator, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FUMAPMS2016
Record Dates: First submitted 2016-11-08; First posted 2016-11-09 (Estimated); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Primary Progressive Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive | interventions — Dimethyl Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active drug (Active Comparator): Dimethyl fumarate, 240mg twice daily for 48 weeks
  Interventions: Drug: Dimethyl fumarate
- Placebo (Placebo Comparator): Placebo Oral Capsules, 2 tablets twice daily for 48 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dimethyl fumarate
  Other Names: Tecfidera; BG-12
  Arms: Active drug
Drug: Placebo — Manufactured to mimic Dimethyl Fumarate capsules
  Arms: Placebo

SUMMARY:
This study aims to evaluate safety and efficacy of dimethyl fumarate treatment in patients with primary progressive multiple sclerosis (PPMS).

Half of the patients will receive dimethyl fumarate and the other half will receive placebo.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a chronic, inflammatory disease of the central nervous system and is presumed to be caused by T cell-mediated autoimmune processes. PPMS has no registered treatment options only symptomatic treatment exists. Progressive forms of MS are characterized clinically by gradual symptom development with or without superimposed relapses.

Fumarates have long been known to have disease-attenuating effects in psoriasis. They have been in routine use in dermatology in Germany for several decades. Dimethyl fumarate has the interesting property of combining immunological effects, at least partly mediated by interference with nuclear factor kappa B and other transcription factors, and also anti-oxidative and neuroprotective effects mediated by activation of the transcription factor Nuclear factor (erythroid-derived 2)-Related Factor 2 (NRF2). Dimethyl fumarate is currently approved for treatment of relapsing-remitting MS by the European medicines Agency in a dose of 240 mg twice per day.

Neurofilament light chain (NFL) is a treatment responsive biomarker of neuronal and axonal death when appearing in the cerebrospinal fluid (CSF) and it has been associated with long-term prognosis in MS. The concentration is often elevated in progressive MS patients. Treatment effect is measured by measuring changes in neurofilament light chain concentration over the course of 48 weeks of treatment with either active drug or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years
* PPMS according to the McDonald (2010) and Lublin (2014) criteria
* Disease duration at least one year
* EDSS ≤ 6.5
* Written informed consent to study participation
* No other signs of significant disease judged by the investigator
* Eligible for randomization to active treatment or placebo as assessed by CSF NFL levels above 380ng/L
* Not eligible for randomization as assessed by CSF biomarker studies but accepts follow-up and open-label treatment per protocol
* Patients not eligible for randomization due to low NFL concentrations in CSF at screening can be followed up after 48 weeks, and are eligible for open-label treatment if they fulfil one of the following clinical criteria of disease progression:
* 1 point increase in EDSS score from screening to week 48 if screening EDSS <6
* 0.5 point increase in EDSS score from screening to week 48 if screening EDSS>5.5
* 2 point increase in a physical functional system
* Worsening in SDMT, 9HPT or T25FW >20% from screening to week 48

Exclusion Criteria:

* Pregnancy or breast feeding
* Lack of effective contraception for women of child-bearing potential
* Relapse within 6 months of inclusion
* Methylprednisolone treatment within 3 months of inclusion
* Treatment with interferon-beta, glatiramer acetate, immunoglobulin G or other immunomodulatory treatment within 6 months of inclusion
* Treatment with mitoxantrone, cyclophosphamide, azathioprine or other immunosuppressive treatment within 6 months of inclusion
* Findings on the screening MRI judged to preclude participation by the treating physician
* Other diseases associated with immunodeficiency
* Other diseases judged to be relevant by the treating physician
* Anticoagulant therapy other than platelet inhibitors
* Active malignant disease in the previous 5 years
* Renal insufficiency or blood creatinine > 150 μmol/l
* Present or chronic infection with hepatitis B virus, hepatitis C virus, HIV (tested in the screening blood samples) or other infections found to be relevant by the treating physician.
* Psychiatric disorders or other disorders impairing the patient's ability to participate in the trial
* Contraindication to MRI
* Known allergy or hypersensitivity to dimethyl fumarate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2019-12-21 (Actual); Study Completion 2020-12-09 (Actual)

PRIMARY OUTCOMES:
Neurofilament light chain in the cerebrospinal fluid (CSF) | 0-48 weeks
  CSF Neurofilament Light Chain (NFL) is measured twice over a course of 48 weeks. Patients will have a spinal tap performed at baseline and again at week 48.

SECONDARY OUTCOMES:
Expanded Disability Status Scale (EDSS) | 0-48 weeks
  We will analyze the difference in EDSS change from screening visit to week 48 between the treatment and placebo group. EDSS is performed by a certified physician, primarily the PI.
Timed 25-Foot Walk (T25FW) | 0-48 weeks
  We will analyze the difference in T25FW change from screening visit to week 48 between the treatment and placebo group. T25FW is evaluated by the principal investigator or a delegated member of the study team.
Nine hole peg test (9HPT) | 0-48 weeks
  We will analyze the difference in 9HPT change from screening visit to week 48 between the treatment and placebo group. 9HPT is evaluated by the principal investigator or a delegated member of the study team.
Symbol digit modalities test (SDMT) | 0-48 weeks
  We will analyze the difference in the SDMT change from screening visit to week 48 between the treatment and placebo group using a general linear model with treatment allocation as factor and the screening SDMT value as covariate. SDMT is evaluated by the principal investigator or a delegated member of the study team.
CSF/Serum Immunoglobulin type G index | 0-48 weeks
  Is assessed from a sample of the cerebrospinal fluid at baseline and at week 48 and change is recorded. The analysis will be performed by the routine diagnostics department at the hospital where the spinal tap is performed.
Cerebrospinal fluid-serum albumin quotient | 0-48 weeks
  We will analyze the difference in change in CSF-serum albumin quotient from screening visit to week 48 between the treatment and placebo group. The analysis will be performed by the routine diagnostics department at the hospital where the spinal tap is performed.
soluble CD14 (sCD14) | 0-48 weeks
  We will analyze the difference in change in sCD14 concentration from screening visit to week 48 between the treatment and placebo group. The analysis is performed by a multiplex luminex assay (R&D systems).
soluble CD27 (sCD27) | 0-48 weeks
  We will analyze the difference in change in sCD27 concentration from screening visit to week 48 between the treatment and placebo group. The analysis is performed by a multiplex luminex assay (R&D systems).
BCMA | 0-48 weeks
  We will analyze the difference in change in BCMA concentration from screening visit to week 48 between the treatment and placebo group. The analysis is performed by a multiplex luminex assay (R&D systems).
Chitinase 3-like-1 | 0-48 weeks
  We will analyze the difference in change in CHI3L1 concentration from screening visit to week 48 visit between the treatment and placebo group. The analysis is performed by a multiplex luminex assay (R&D systems).
Myelin Basic protein (MBP) | 0-48 weeks
  We will analyze the difference in change in MBP concentration from screening visit to week 48 between the treatment and placebo group. The analysis is performed by a enzyme-linked immunosorbent assay (ELISA) (R&D DuoSet).
Number of new or enlarged T2 lesions | 0-48 weeks
  We will analyze the number of new or enlarging T2 lesions from screening visit to W48 between the treatment and placebo group. This analysis will be performed by our collaborator at Hvidovre Hospital (Danish Research Center for Magentic Resonance)
Fractional anisotropy (FA) in Normal Appearing White Matter (NAWM) | 0-48 weeks
  We will analyze the difference in change from screening to W48 of FA in NAWM between the treatment and placebo group. This analysis will be performed by our collaborator at Hvidovre Hospital (Danish Research Center for Magentic Resonance)
Change in lesion volume | 0-48 weeks
  We will analyze the change from screening to W48 in lesion volume. This analysis will be performed by our collaborator at Hvidovre Hospital (Danish Research Center for Magentic Resonance)
Change from screening in in magnetization transfer ratio (MTR) of T2 lesions | 0-48 weeks
  We will analyze the difference in change from screening to W48 in MTR of T2 lesions between the treatment and placebo group. This analysis will be performed by our collaborator at Hvidovre Hospital (Danish Research Center for Magentic Resonance).
Thalamic volume | 0-48 weeks
  We will analyze the difference in change from screening to W48 of thalamic volume between the treatment and placebo group. This analysis will be performed by our collaborator at Hvidovre Hospital (Danish Research Center for Magentic Resonance).
Percent brain volume change (PBVC) | 0-48 weeks
  We will analyze the difference in percentage change in brain volume from screening visit to week 48 between the treatment and placebo group. This analysis will be performed by our collaborator at Hvidovre Hospital (Danish Research Center for Magentic Resonance).

OTHER OUTCOMES:
BVMTR | 0-48 weeks & 48-96 weeks
  Change from screening for Brief Visuospatial Memory Test Revised (BVMTR) The test is performed by the principal investigator or a delegated member of the study team.
California Verbal Learning Test 2 (CVLT-II) | 0-48 weeks & 48-96 weeks
  Change from screening for California Verbal Learning Test 2 (CVLT-II). The test is performed by the principal investigator or a delegated member of the study team.
UDI | 0-48 weeks & 48-96 weeks
  The questionnaire is handed out at screening visit, week 48 and week 96.
FSMC | 0-48 weeks & 48-96 weeks
  The questionnaire is handed out at screening visit, week 48 and week 96.
MSIS-29 | 0-48 weeks & 48-96 weeks
  The questionnaire is handed out at screening visit, week 48 and week 96.
Number of Gadolinium (Gd) enhancing lesions on MRI | 0-48 weeks & 48-96 weeks
  Change from screening/W48 in number of Gd-enhancing lesions.
Number of new T2 lesions | 48-96 weeks
  Change from screening in number of new T2 lesions
Number of enlarged T2 lesions | 48-96 weeks
  Change from screening in number of enlarged T2 lesions
Brain volume change | 0-48 weeks & 48-96 weeks
  Change from screening/W48 in volume of cortical grey matter (CGM), normal appearing white matter (NAWM), thalamus, putamen and lesion volume.
Change in Magnetization Transfer Ratio (MTR). | 0-48 weeks & 48-96 weeks
  Change from screening/W48 in Magnetization Transfer Ratio (MTR) of CGM, NAWM, the putamen and thalamic nuclei
Change in diffusion tensor imaging (DTI) measures (FA and mean diffusivity). | 0-48 weeks & 48-96 weeks
  Change from screening/W48 in diffusion tensor imaging (DTI) measures (FA and mean diffusivity) of CGM, NAWM (except FA in NAWM from screening to week 48), lesions, the putamen and thalamic nuclei.
Cross sectional area at C2 level of the cervical spinal cord on MRI | 0-48 weeks & 48-96 weeks
  Change from screening/W48 in the cross sectional area at the C2 level of the cervical spinal cord on MRI.
Circle drawing test at the time of the MRI | 0-48 weeks & 48-96 weeks
  At the time of MRI (screening, week 48 and week 96) a circle drawing test will be performed.
Change in Serum Neurofilament Light Chain (serum NFL) | 0-48 weeks & 48-96 weeks
  Is assessed from a blood sample at screening visit, W48 visit, and W96 visit. The analysis is performed by the neuroimmunology laboratory with a commercially available SIMOA-assay (Quanterix).

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Lando Talbot, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Danish Multiple Sclerosis Center, Department of neurology, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] von Essen MR, Talbot J, Hansen RHH, Chow HH, Lundell H, Siebner HR, Sellebjerg F. Intrathecal CD8+CD20+ T Cells in Primary Progressive Multiple Sclerosis. Neurol Neuroimmunol Neuroinflamm. 2023 Jun 27;10(5):e200140. doi: 10.1212/NXI.0000000000200140. Print 2023 Sep. PMID 37369602
- [Derived] Hojsgaard Chow H, Talbot J, Lundell H, Gobel Madsen C, Marstrand L, Lange T, Mahler MR, Buhelt S, Holm Hansen R, Blinkenberg M, Romme Christensen J, Soelberg Sorensen P, Rode von Essen M, Siebner HR, Sellebjerg F. Dimethyl Fumarate Treatment in Patients With Primary Progressive Multiple Sclerosis: A Randomized, Controlled Trial. Neurol Neuroimmunol Neuroinflamm. 2021 Aug 24;8(5):e1037. doi: 10.1212/NXI.0000000000001037. Print 2021 Sep. PMID 34429340

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-28): https://cdn.clinicaltrials.gov/large-docs/58/NCT02959658/Prot_SAP_000.pdf